CLINICAL TRIAL: NCT04409145
Title: Open-Label, Intra Subject, Dose Escalation (Part 1) Followed by Randomized, Double Blind, Placebo Controlled (Part 2) Trial of Topical VT30 in Pts With Venous, Lymphatic or Mixed Malformations Associated With PIK3CA or TEK Genetic Mutations
Brief Title: First in Human Trial of Topical VT30 in Pts With Venous/Lymphatic Malformations Assoc With PIK3CA or TEK Gene Mutations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Part 1 complete; Part 2 will not be completed.
Sponsor: Venthera, Inc., a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VT30-101
Record Dates: First submitted 2020-05-11; First posted 2020-06-01 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Venous Malformation; Lymphatic Malformation; Venolymphatic Malformation
MeSH Terms: conditions — Lymphatic Abnormalities

STUDY DESIGN:
Intervention Model Description: Part 1: Open-label, 4-sequence, escalating repeat-application cohort study, with intra-subject and inter-cohort dose escalation to determine safety and tolerability, and maximum feasible dose/maximum tolerable dose Part 2: Randomized, placebo-controlled, double-blind, safety and exploratory efficacy study
Masking Description: Part 1: Open label Part 2: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VT30 (Experimental): VT30 is a PI3K-inhibitor prodrug, formulated as a topical gel and dispensed from a metered dose pump; administration is once or twice daily, applied to target-treatment area(s) on the skin. One pump action dispenses 250 µL of gel, intended to treat an area of 140 cm2.
  Interventions: Drug: VT30

INTERVENTIONS:
Drug: VT30 — VT30 gel is intended as a topical treatment of cutaneous VMs, LMs, or VLMs that driven by inappropriate PI3K activation. In the skin, VT30 is rapidly metabolized to VT10, an active drug form, and is intended to sufficiently permeate the stratum corneum and achieve target engagement. It is expected that VT30 will lead to amelioration of the signs and symptoms of cutaneous VMs, LMs and/or VLMs.

SUMMARY:
VT30-101 is a 2-part first-in-human trial of topically administered VT30 to subjects with cutaneous venous malformations, lymphatic malformations, or mixed venolymphatic malformations associated with PIK3CA or TEK mutations.

Part 1 is a 4-week treatment, open-label, 4-sequence, escalating repeat-application cohort study, with intra-subject and inter-cohort dose escalation.

Part 2 is a 12-week treatment, randomized, placebo-controlled, double-blind, safety and exploratory efficacy study. Part 2 will be initiated only after the successful completion of Part 1 with results that demonstrate the general safety and tolerability of topically applied VT30. Up to 12 subjects who complete Part 1 may be enrolled into Part 2 of the study.

The primary objective is to evaluate the safety and tolerability of VT30. The study will also determine the dose and regimen of VT30 to be carried into Part 2 of the protocol. Other aims include documenting plasma drug levels of VT30 and VT10 and, on an exploratory basis, examining pharmacologic target engagement and change in potential efficacy readouts.

DETAILED DESCRIPTION:
VT30-101 is designed as a Phase 1/2, first-in-human study of topically administered VT30 to subjects with cutaneous venous malformations (VMs), lymphatic malformations (LMs), or mixed venolymphatic malformations (VLMs) associated with phosphatidylinositol 3-kinase catalytic alpha polypeptide (PIK3CA) or tyrosine receptor kinase (TEK) mutations. Capillary involvement and/or extension of the lesion into subcutaneous tissues is permitted.

The study will occur in 2 parts, and in both study parts, subjects will participate in a Screening Period (up to 6 weeks) before beginning the indicated Treatment Period.

Part 1 will be an open-label, 4-sequence, escalating repeat-application study comprised of up to 4 cohorts (3 subjects per cohort, with 3 up to 6 in Cohort 4, or the final Part 1 cohort). In each cohort, subjects will be given topical VT30 for a 4-week Treatment Period. Subjects will begin treatment with the designated dose on Day 1. After 2 weeks, the Investigator will examine the treated surface area and determine if the formulation is tolerated such that the subject may apply the next dose strength of VT30 gel for the remaining duration of the Treatment Period.

Specifically, the following gel dose strengths (concentrations) are planned for Cohorts 1 through 3 in Part 1:

* Cohort 1: initiate dosing with 0.12% (w/w) gel and progress to 0.6% (w/w) gel for the final 2 weeks of the Part 1 Treatment Period (if the lower dose is tolerated)
* Cohort 2: initiate dosing with 0.6% (w/w) gel and progress to 1.2% (w/w) gel for the final 2 weeks of the Part 1 Treatment Period (if the lower dose is tolerated)
* Cohort 3: initiate dosing with 1.2% (w/w) gel and progress to 2.3% (w/w) gel for the final 2 weeks of the Part 1 Treatment Period (if the lower dose is tolerated)

A Safety Review Committee (SRC), with sponsor, investigator and independent medical representation, will provide oversight and guidance for study conduct. After 3 subjects have been dosed for at least 21 days in any of the first three Part 1 cohorts, the SRC may request additional data, approve initiation of the subsequent cohort, or mandate that additional subjects to be enrolled at either the higher or lower dose within the cohort.

After 9 subjects in Cohorts 1 through 3 (3 subjects per cohort) have completed the 4-week Treatment Period, the SRC will determine if additional subjects should be assigned to Cohort 4 (or the final Part 1 cohort) to receive the MTD (maximum tolerated dose) or MFD (maximum feasible dose) strength of VT30. Subjects in Cohort 4 will receive the designated dose strength and regimen of VT30 for a full 4 weeks.

Following the completion of Cohort 4 in Part 1, the SRC will determine whether to authorize initiation of Part 2 and will confirm the dose level and regimen to be administered in Part 2.

Part 2 will be a randomized, placebo-controlled, double-blind study containing 36 subjects assigned in a 2:1 ratio to receive either VT30 or placebo. Up to 12 subjects who complete Part 1 may enroll in Part 2, provided they meet all Part 2-specific inclusion criteria with no applicable exclusions.

After the first 12 subjects in Part 2 have completed 4 weeks of treatment, the SRC will conduct a review of blinded safety data to confirm no revisions or changes are needed to the protocol. Subsequent reviews may also be conducted to ensure continued acceptable safety and tolerability.

After subjects complete their designated Treatment Period (in Part 1 or Part 2), they will participate in a 4-week post treatment Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed the current approved informed consent form
2. Have a clinically or phenotypically defined VM, LM, or mixed VLM affecting the skin
3. Lesion genotyping confirms either PIK3CA or TEK mutations, known to be pathogenic
4. Agrees to use contraception if of childbearing potential
5. Be willing and able to comply with the protocol and be available for the entire study
6. Be at least 18 to 60 years of age
7. Lesion must be amenable to defining a contiguous study treatment area of 140 cm2

Exclusion Criteria:

1. Lesion to be treated is on the face or involves mucosa
2. Presence of ulcerations on the target-treatment lesion
3. Known systemic hypersensitivity to the VT30 drug substance, its inactive ingredients, or the vehicle
4. Uncontrolled diabetes mellitus
5. Hyperlipidemia that is poorly controlled on current treatment
6. Pregnant or nursing, planning to become pregnant, or planning to father a child during the study
7. History of malignancy except successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix
8. Major surgery within 8 weeks of Screening, or a surgical, laser or other procedure involving the target lesion within 8 weeks of Screening, or planned to occur during the study
9. Any other medical or personal condition that, in the opinion of the Investigator, may potentially compromise the safety or compliance of the subject, or may preclude the subject's successful completion of the clinical study
10. Medically significant infection (eg, cellulitis or abscess, or a systemic infection) within 8 weeks of Screening
11. Ongoing therapy with another topical treatment or any medication that inhibits PI3K, Akt pathway, or the mTOR pathway, or in the opinion of the Investigator, the subject requires systemic therapy for their vascular malformation condition
12. Use of a biologic or systemic immunosuppressive agent within 3 months of Screening
13. Systemic use of corticosteroids, within 30 days of Screening
14. Treatment with a small molecule investigational product within 30 days of Screening, or with any investigational biologic products within 3 months of Screening
15. Positive for hepatitis C antibody, hepatitis B surface antigen, hepatitis B core antibody, or human immunodeficiency virus
16. Alanine transaminase or aspartate transaminase laboratory values in excess of 1.5X the upper limit of normal at Screening
17. Hemoglobin A1c is >8%
18. Any other clinically significant laboratory or testing abnormality that, in the opinion of the Investigator, might confound the study, interfere with the subject's ability to complete the study, or represent a meaningful safety risk upon study enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability | From pre-treatment to 4 weeks of treatment
  Composite of adverse events and changes in physical exam findings, vital signs, lab tests, and electrocardiogram evaluations

SECONDARY OUTCOMES:
Maximum feasible dose / maximum tolerable dose | From pre-treatment to 4 weeks
  The MTD or MFD strength will be determined based on results from Part 1, and will inform the dose strength to be used in Part 2
Tissue and serum drug levels | From pre-treatment to 4 weeks
  Plasma levels of VT30 and VT10 will be assessed following topical administration of VT30 to determine level of systemic exposure

OTHER OUTCOMES:
Maximum tissue concentration of study drug | From pre-treatment to 4 weeks
  As assessed by treated lesion tissue levels of phosphoproteins, as an indicator of local target engagement
Changes in Pain | From pre-treatment to 4 weeks
  Assessed by subjects' self-reporting their pain, related to the treated lesion, on a Numerical Rating Scale
Changes in lesion | From pre-treatment to 4 weeks
  Assessed by change in appearance of the treated lesion
Changes in management of lesion bleeding, oozing, or discharge | From pre-treatment to 4 weeks
  Assessed by subject-reported difficulty managing bleeding, oozing, or discharge from the treated lesion

CONTACTS AND LOCATIONS:
Overall Officials: Michael Henderson, Study Director — Venthera, Inc., a BridgeBio company
Locations (15):
- United States (15):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital/UAMS, Little Rock, Arkansas
  - Stanford University Medical Center, Palo Alto, California
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, San Diego, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Indiana University Health (Riley Children's Hospital and University Hospital), Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Raleigh, North Carolina
  - Cincinnatti Children's Hospital, Cincinnati, Ohio
  - University Hospitals- Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - University of Virginia Department of Dermatology, Charlottesville, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No